CLINICAL TRIAL: NCT02728778
Title: Botulinum Toxin A for Emotional Stabilization in Borderline Personality Disorder (BPD)
Acronym: BTX-BPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Prof. Dr. Tillmann Krüger, M.D., Associate Professor, Hannover Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: V4.11-BTX-BPD
Record Dates: First submitted 2016-03-31; First posted 2016-04-05 (Estimated); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Botulinum Toxins, Type A; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum toxin A (Active Comparator): Single administration of incobotulinumtoxin A into the forehead (glabellar region); 34 U in five injection sites.
  Interventions: Drug: incobotulinumtoxin A
- Acupuncture (Other): Patients will receive four facial acupuncture treatments every two weeks.
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Drug: incobotulinumtoxin A — Application of botulinum toxin A into the forehead
  Other Names: Botox
  Arms: Botulinum toxin A
Procedure: Acupuncture — Application of acupuncture into the forehead
  Arms: Acupuncture

SUMMARY:
The main objective of the trial is to test whether a single application of botulinum toxin A into the glabellar region will lead to emotional stabilization in borderline personality disorder through paralysis of facial muscles/attenuation of negative emotions.

DETAILED DESCRIPTION:
Afferent feedback from facial muscles is believed to enhance emotional states (facial feedback theory). The facial expression of negative emotions involves facial muscles of the glabellar region. It has been shown that paralysis of facial muscles in the forehead using botulinum toxin A leads to the improvement of depressive symptoms. It is believed that the limited ability to express these emotions alleviates depressive symptoms. As Borderline personality disorder is characterized by negative emotions expressed via facial muscles in the forehead, it is hypothesized that BPD patients could profit from botulinum toxin treatment.

ELIGIBILITY:
Inclusion Criteria:

1. female
2. 18-40 years
3. diagnosed BPD according to ICD-10 (F60.31) and SKID II
4. stable treatment
5. mastery of the German language
6. effective contraception
7. willingness to and acceptance of treatment with either botulinum toxin A or acupuncture

Exclusion Criteria:

1. Comorbid disorders of all ICD-10 groups o F0,

   * F1 (with exception of F1x.1),
   * F2,
   * F3 (with exception of 32.0 and F33.0),
   * F7 and disorders essentially defining the clinical picture from sections
   * F4,
   * F5,
   * F6.
2. Contraindication for treatment with botulinum toxin A according to the IMP's SmPC (e.g. myasthenia gravis, Lambert Eaton-syndrome or other impairments in neuromuscular function)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Zanarini Scale for Borderline personality disorder (ZAN-BPD) | 8 weeks
  BPD severity measure expert rating

SECONDARY OUTCOMES:
Borderline symptom list (BSL-23) | 4, 8 and 16 weeks
  BPD severity measure self rating
Montgomery-Asberg-Depression-Rating-Scale (MADRS) | 4, 8 and 16 weeks
  depression severity measure expert rating
Beck Depression Inventory (BDI) | 4, 8 and 16 weeks
  depression severity measure self rating

CONTACTS AND LOCATIONS:
Overall Officials: HCTC, Study Chair — Hannover Clinical Trial Center HCTC GmbH
Locations (2):
- Germany (2):
  - Hannover Medical School, Hanover, Lower Saxony
  - Asklepios Klinik Nord-Ochsenzoll, Hamburg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wollmer MA, Neumann I, Jung S, Bechinie A, Herrmann J, Muller A, Wohlmuth P, Fournier-Kaiser L, Sperling C, Peters L, Kneer J, Engel J, Jurgensen F, Schulze J, Nagel M, Prager W, Sinke C, Kahl KG, Karst M, Dulz B, Kruger THC. Clinical effects of glabellar botulinum toxin injections on borderline personality disorder: A randomized controlled trial. J Psychopharmacol. 2022 Feb;36(2):159-169. doi: 10.1177/02698811211069108. Epub 2022 Feb 1. PMID 35102782